CLINICAL TRIAL: NCT04830098
Title: Comparison of the Effectiveness of Spinal Stabilization Exercises and Chiropractic Spinal Manipulation in Healthy Individuals
Brief Title: Comparison of the Effectiveness of Spinal Stabilization Exercises and Chiropractic Spinal Manipulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Mesut Arslan, Head of Therapy and Rehabilitation Department, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHRİOEXERCİSE001
Record Dates: First submitted 2021-03-26; First posted 2021-04-02 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-04

CONDITIONS: Healthy Individuals
Keywords: Spinal stabilization; Exercise; Manipulation; Chiropractic
MeSH Terms: conditions — Motor Activity | interventions — Manipulation, Chiropractic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stabilization group (Experimental): Stabilization group will be given stabilization exercises for a total of 18 sessions, 3 times a week for 6 weeks, each session for 45 minutes.
  Interventions: Other: Spinal stabilization exercises
- Manipulation group (Experimental): Manipulation group be applied high-speed low-amplitude (HVLA) chiropractic manipulation for a total of 6 sessions, once a week for 6 weeks.
  Interventions: Other: Chiropractic manipulation
- Stabilization and Manipulation group (Experimental): Stabilization and Manipulation group will be given both stabilization exercises and manipulation exercises.
  Interventions: Other: Spinal stabilization exercises; Other: Chiropractic manipulation
- Control group (No Intervention): No application will be made in the control group.

INTERVENTIONS:
Other: Spinal stabilization exercises — It will be given stabilization exercises for a total of 18 sessions, 3 times a week for 6 weeks, each session for 45 minutes.
  Arms: Stabilization and Manipulation group; Stabilization group
Other: Chiropractic manipulation — It will be applied high-speed low-amplitude (HVLA) chiropractic manipulation for a total of 6 sessions, once a week for 6 weeks.
  Arms: Manipulation group; Stabilization and Manipulation group

SUMMARY:
It is the study of the effectiveness of spinal stabilization exercises and chiropractic spinal manipulation in healthy individuals.

In addition, it was planned to investigate the effects of spinal stabilization exercises and manipulation on muscle strength, muscular endurance, balance and proprioception, depression and quality of life.

DETAILED DESCRIPTION:
It is the study of the effectiveness of spinal stabilization exercises and chiropractic spinal manipulation in healthy individuals.

In addition, it was planned to investigate the effects of spinal stabilization exercises and manipulation on muscle strength, muscular endurance, balance and proprioception, depression and quality of life.

Eighty healthy individuals between the ages of 18-45 who voluntarily participated in the study from students or academic/administrative staff at Gümüşhane University were included in the study. The study program was explained to the participants in line with the Informed Consent Form. It was included in the study after the relevant form was signed by the participant.

Healthy individuals to participate in the study will be randomly divided into 4 groups; randomization will be done by "Research Randomizer" computer program. Group 1 Stabilization group (n = 20), Group 2 Manipulation group (n = 20), Group 3 Stabilization and Manipulation group (n = 20), Group 4 Control group (n = 20). Group 1 will be given stabilization exercises for a total of 18 sessions, 3 times a week for 6 weeks, each session for 45 minutes. Group 2 will be applied high-speed low-amplitude (HVLA) chiropractic manipulation for a total of 6 sessions, once a week for 6 weeks. Group 3 will be given both stabilization exercises and manipulation exercises. The fourth group will be followed as a control group and no application will be made. Prone plunk, side plunk and sorenson tests for muscular endurance in the individuals participating in the study; Quadriceps muscle strength for muscle strength assessment; Joint position sense for propioception; Y balance test for balance; Short Form-36 (SF-36) for quality of life; Beck Depression Inventory was planned to be evaluated before, after and 1 months for psychosomatic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer individuals (Female and Male),
* Between the ages of 18-45,
* No pain, trauma or surgery history in the last 6 months,
* Without any chronic disease (Obesity, Diabetes, Hypertension, Osteoporosis),
* Individuals who had not received any treatment for spinal problems before were included in the study.

Exclusion Criteria:

* Conditions where chiropractic spinal manipulation is contraindicated (Inflammation, infection, malignancy, blood coagulation disorder, etc.)
* Any injury during the working process,
* Individuals who did not attend the work program regularly were not included in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Joint position sense change | Before starting study, after the study is finished, 1 month after the end of the study
  The knee to be evaluated in a closed and quiet environment was positioned at 60 degrees of flexion joint angle for five seconds, and the person was asked to perceive this angular position. Then, the knee was relaxed and the person was asked to return to the joint position he perceived and hold for five seconds at that point. The difference is considered as the error angle. The error angle was calculated by taking the average of 3 trials. Measurements were made with the participants' eyes closed
Quadriceps muscle strength change | Before starting study, after the study is finished, 1 month after the end of the study
  During the test, after the participant completed the maximum knee extension, the evaluator stabilized the applied thigh with one hand and placed the dynamometer perpendicular to the leg 1-2 cm above the level of the malleoli with the other hand. A thin towel was placed between the dynamometer and the leg so that the dynamometer did not hurt the leg during the measurement. During the test, the "make test" technique, which requires isometric contraction, was applied. (Make test is the protocol of the person applying the maximum force against the device while the meter keeps the dynamometer constant). After the knee extension was completed, the participant was asked to maintain the maximum isometric contraction for 5 seconds. The average of 3 consecutive maximum contraction measurement values made at 30-second intervals was calculated
Y balance test change | Before starting study, after the study is finished, 1 month after the end of the study
  It was used for dynamic balance of individuals. The validity reliability of the test was determined by Plisky et al. ICC range was 0.85-0.01 intrarater and 0.99-1.00 interrater [30]. The amount of lying on the dominant extremities of the individuals was measured. The subject was asked to stand on one foot at the midpoint of the test setup and touch with the tip of the toe while maintaining his balance with the other foot in the anterior, posteromedial and posterolateral directions. The test was repeated 3 times in all directions, averaged and recorded in cm.
Prone Plank Test change | Before starting study, after the study is finished, 1 month after the end of the study
  It is a valid and reliable test used to measure the endurance of core region muscles [27]. The participant is asked to lie face down and rise on their elbows and toes while keeping the body in a straight line. The total time is recorded. The time is stopped if the participant lowers or lifts his body.
Side Plank Test change | Before starting study, after the study is finished, 1 month after the end of the study
  It evaluates the endurance of the lateral trunk flexor muscles. The participant is asked to lie on his side on the elbow with the legs in full extension. Participant is asked to lift the lower limbs so that the hips and back are aligned and maintain this position. The total time is recorded. If the participant dropped his hip, the time was stopped. Measurements were repeated on both sides, right and left.
Sorenson test change | Before starting study, after the study is finished, 1 month after the end of the study
  Participant lies face down with his torso hanging from the table above the Anterior Superior Iliac Spine (ASIS) level. Thighs and legs are stabilized using straps. Participant then places his hands diagonally on the shoulders and is asked to lift his body at the same level with the table. Participant is asked to hold this position as long as possible and the total time is recorded.

SECONDARY OUTCOMES:
Short Form-36 change | Before starting study, after the study is finished, 1 month after the end of the study
  Developed to evaluate the quality of life, this scale was developed by Koçyiğit et al. Turkish validity and reliability study was conducted by [33]. SF-36 is a 36-item scale that includes physical and mental health inquiries. The high score obtained from the scale, which is evaluated between 0 and 100 points, indicates good health.
Beck Depression Inventory change | Before starting study, after the study is finished, 1 month after the end of the study
  Hisli et al. It is a scale consisting of 21 items, whose Turkish validity and reliability study was conducted by [35]. The high score obtained from the scale, which is between 0 and 63 points, indicates the presence of high depression. 0-9 points are defined as minimal depression, 10-16 points mild depression, 17-29 points moderate depression, and 30-63 points severe depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Gumushane University, Gümüşhane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No